CLINICAL TRIAL: NCT05199103
Title: Single-centre, Safety and Efficacy, Open-label Study Evaluating Antithymocyte Globulin Treatment in Subjects With Graves Orbitopathy
Brief Title: Antithymocyte Globulin as a Second Line Therapy in Graves Orbitopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Gabriela Handzlik, Principal Investigator, Medical University of Silesia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNW-1-075/N/8/K
Record Dates: First submitted 2021-12-27; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Graves Orbitopathy
Keywords: Graves disease; proptosis; antithymocyte globulin
MeSH Terms: conditions — Graves Ophthalmopathy; Graves Disease; Exophthalmos | interventions — Antilymphocyte Serum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rabbit antithymocyte globulin (rATG) (Experimental)
  Interventions: Drug: rabbit anti-thymocyte globulin

INTERVENTIONS:
Drug: rabbit anti-thymocyte globulin — 0.8 - 1.0 mg/kg of rATG (cumulative dose of 150-200 mg given intravenously in two or three divided doses, 24 hours apart) after premedication with methylprednisolone i.v. (in total dose of 375 mg), 1 mg of antihistaminic agent clemastine and 1000 mg paracetamol i.v.

SUMMARY:
The overall objective of the study is to evaluate the safety and efficacy of rabbit antithymocyte globulin in the treatment of Graves orbitopathy (GO) after ineffective treatment with moderate-to-high doses of glucocorticoids.

DETAILED DESCRIPTION:
This is a prospective interventional, single-center study examining the safety and efficacy of rabbit antithymocyte globulin (rATG) in adult patients with active moderate-to-severe GO after ineffective treatment with moderate-to-high doses of glucocorticoids. All enrolled participants will receive 0.8 - 1.0 mg/kg of rATG (cumulative dose of 150-200 mg given intravenously in two or three divided doses, 24 hours apart) after premedication with methylprednisolone i.v. (in total dose of 375 mg), 1 mg of antihistaminic agent clemastine and 1000 mg paracetamol i.v.

In order to assess efficacy and safety of the treatment, patients will be evaluated at baseline and at 6, 12, 24 and 48 weeks. Baseline and subsequent evaluation will involve medical history, physical examination, including detailed eye examination, laboratory assessment (thyroid-stimulating hormone [TSH], flow cytometry, TSH-receptor antibodies, CBC) and orbital magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Graves' disease associated with active thyroid eye disease and a clinical activity score of ≥ 3
* Euthyroid or with mild hypo- or hyperthyroidism defined as free thyroxine (FT4) and free triiodothyronine (FT3) levels less than 50% above or below the normal limits
* previous ineffective treatment (partial response, recurrence or progression of symptoms) with moderate-to-high doses of glucocorticoids (at least 4.5 g of methylprednisolone)

Exclusion Criteria:

* hypersensitivity to rabbit proteins or to any product excipients
* active acute or chronic infections
* latent tuberculosis
* leucopenia below 3000/μl
* lymphopenia below 400/μl
* thrombocytopenia below 75000/μl
* coagulation disorders
* active malignancy and pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
≥2 point change in Clinical Activity Score from baseline | Week 6, 12, 24, 48
change in proptosis | 48 weeks
a diplopia response | 48 weeks
change of distant best-corrected visual acuity | Week 6, 12, 24, 48
change of mean retinal sensitivity | Week 6, 12, 24, 48

SECONDARY OUTCOMES:
changes in CD4/CD8 ratio | Week 6, 12, 24, 48
changes in TSH-receptor antibodies level | Week 6, 12, 24, 48
increase in 1 degree amplitude in Pattern visual evoked potential (VEP) by 1 µV | Week 6, 12, 24, 48

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Chudek, Prof., Principal Investigator — Medical University of Silesia
Locations (1):
- Department of Internal Medicine and Oncological Chemotherapy, Medical Faculty in Katowice, Medical University of Silesia, Katowice, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarnat-Kucharczyk M, Swierkot M, Handzlik G, Kulawik G, Jagoda K, Grochola-Malecka I, Fryzewska J, Mrukwa-Kominek E, Chudek J. Antithymocyte Globulin as Second-Line Therapy in Graves Orbitopathy-Preliminary Results From a Prospective Single-Center Study. Front Endocrinol (Lausanne). 2022 May 9;13:871009. doi: 10.3389/fendo.2022.871009. eCollection 2022. PMID 35615718